CLINICAL TRIAL: NCT05428007
Title: A Phase II Study of the Interleukin-6 Receptor Inhibitor Sarilumab in Combination With Ipilimumab, Nivolumab and Relatlimab in Patients With Unresectable Stage III or Stage IV Melanoma
Brief Title: Interleukin-6 Receptor Inhibitor Sarilumab in Combination With Ipilimumab, Nivolumab and Relatlimab in Patients With Unresectable Stage III or Stage IV Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-00325
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Melanoma; Unresectable Melanoma
MeSH Terms: conditions — Melanoma | interventions — sarilumab; Ipilimumab; CTLA-4 Antigen; Nivolumab; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Stage I: sarilumab, ipilimumab, nivolumab and relatlimab (Experimental): Participants with unresectable Stage III/Stage IV melanoma receive sarilumab at 150 mg flat dose is administered subcutaneously every 2 weeks for 12 doses from day 1, cycle 1 in combination with a regimen of ipilimumab at 1 mg/kg every 8 weeks and fixed dose nivolumab at 480 mg and relatlimab at 160 mg flat dose every 4 weeks two times during the 8-week induction period, then the same regimen again up to week 16, and up to week 24 in maintenance. After week 24 the regimen will be ipilimumab at 1 mg/kg every 8 weeks and fixed dose nivolumab at 480 mg with relatlimab at 160 mg flat dose every 4 weeks for 8 week cycles for up to a total of 2 years.
  Interventions: Drug: Sarilumab; Drug: Ipilimumab Injection; Drug: Nivolumab/Relatlimab
- Stage II: ipilimumab, nivolumab and relatlimab (Experimental): Participants with unresectable Stage III/Stage IV melanoma receive a regimen of ipilimumab at 1 mg/kg every 8 weeks and fixed dose nivolumab at 480 mg and relatlimab at 160 mg flat dose every 4 weeks two times during the 8-week induction period, then the same regimen again up to week 16, and up to week 24 in maintenance. After week 24 the regimen will be ipilimumab at 1 mg/kg every 8 weeks and fixed dose nivolumab at 480 mg with relatlimab at 160 mg flat dose every 4 weeks for 8 week cycles for up to a total of 2 years.
  Interventions: Drug: Ipilimumab Injection; Drug: Nivolumab/Relatlimab
- Stage II: sarilumab, ipilimumab, nivolumab and relatlimab (Experimental): Participants with unresectable Stage III/Stage IV melanoma receive sarilumab at 150 mg flat dose is administered subcutaneously every 2 weeks for 12 doses from day 1, cycle 1 in combination with a regimen of ipilimumab at 1 mg/kg every 8 weeks and fixed dose nivolumab at 480 mg and relatlimab at 160 mg flat dose every 4 weeks two times during the 8-week induction period, then the same regimen again up to week 16, and up to week 24 in maintenance. After week 24 the regimen will be ipilimumab at 1 mg/kg every 8 weeks and fixed dose nivolumab at 480 mg with relatlimab at 160 mg flat dose every 4 weeks for 8 week cycles for up to a total of 2 years.
  Interventions: Drug: Sarilumab; Drug: Ipilimumab Injection; Drug: Nivolumab/Relatlimab

INTERVENTIONS:
Drug: Sarilumab — Injectable solutions of sarilumab are formulated in 2 mL of aqueous solution in a 5 mL vial containing 175 mg/ml of sarilumab arginine (8.94 mg), histidine (3.71 mg), polysorbate 20 (2.28 mg), sucrose (57 mg) and Water for Injection USP.Patients will be administered sarilumab at a dose of 150 mg subcutaneously in combination with ipilimumab, nivolumab and relatlimab given intravenously, with nivolumab/relatlimab given intravenously, or sarilumab at a dose of 150 mg subcutaneously given alone.
  Other Names: REGN88
  Arms: Stage I: sarilumab, ipilimumab, nivolumab and relatlimab; Stage II: sarilumab, ipilimumab, nivolumab and relatlimab
Drug: Ipilimumab Injection — Ipilimumab injection is a sterile, nonpyrogenic, clear to slightly opalescent, colorless to pale yellow solution, single-use, preservative-free, isotonic aqueous solution that may contain particles. It is formulated at a concentration of 5 mg/mL ipilimumab in TRIS hydrochloride (also known as 2-amino-2-hydroxymethyl-1,3-propanediol hydrochloride), sodium chloride, mannitol, pentetic acid (also known as diethylenetriaminepentaacetic acid or DTPA), polysorbate 80, and water at pH 7.0. Sodium hydroxide and/or hydrochloric acid may be used to adjust the pH of the solution. Ipilimumab Injection 200 mg/40 mL (5 mg/mL) is packaged in a 50-cc Type I flint molded glass vials.
  Other Names: BMS-734016; MDX010; MDX-CTLA4
Drug: Nivolumab/Relatlimab — The FDC drug product, referred to as nivolumab/relatlimab, contains relatlimab and nivolumab in a single vial in a kit of 2 vials. The product is a sterile, non-pyrogenic, single-use, isotonic aqueous solution for IV infusion. It is formulated at a total protein concentration of 16 mg/mL (4 mg/mL relatlimab and 12 mg/mL nivolumab) and is packaged in a 20-cc glass vial in a kit of two vials. Each vial contains 80 mg of relatlimab and 240 mg of nivolumab.
  Other Names: BMS-986213

SUMMARY:
This study will evaluate how safe the study drug is, how well patients tolerate it, how it works in the body, and the disease's response to the drug. The study drug being tested is sarilumab, when given with the combination of ipilimumab, nivolumab, and relatlimab in patients like yourself, with stage III or stage IV melanoma that cannot be removed by surgery. Previous studies have provided a strong rationale for combining sarilumab, with ipilimumab, nivolumab and relatlimab in metastatic melanoma to reduce side effects and potentially work better for your type of cancer. Sarilumab is an FDA-approved inhibitor of the receptor for the cytokine IL-6, currently approved for the treatment of rheumatoid arthritis, but it is not FDA-approved to treat melanoma. This means that the use of Sarilumab to treat melanoma is considered investigational. The other drugs which will be administered in this study, ipilimumab and nivolumab, are also monoclonal antibodies, but they target different proteins. Ipilimumab and nivolumab are both approved by the FDA to treat advanced stage III and IV melanomas. The nivolumab + relatlimab FDC (fixed dose combination) being used in this study is considered investigational, meaning it is not approved by the FDA. The combination of sarilumab, ipilimumab, nivolumab and relatlimab is considered investigational because it has not yet been approved by the FDA. The FDA has given its permission to study the investigational combination of these drugs in this research study.

DETAILED DESCRIPTION:
This is a Phase II study conducted in two stages. In the first stage, up to 33 patients will be treated with all four drugs in a single arm open label trial. In the second stage, 72 patients will be randomized 1:1 to receive ipilimumab, nivolumab and relatlimab with or without sarilumab for up to 24 weeks. The study will include an assessment of the safety and tolerability and overall response rates of sarilumab administered concurrently at 150 mg flat dose every 2 weeks for 12 doses in combination with ipilimumab for three doses given every 8 weeks, and fixed dose nivolumab and relatlimab given every 4 weeks for six doses to week 24, then maintenance nivolumab and relatlimab every 4 weeks and ipilimumab every 8 weeks for up to a total of two years to patients with advanced melanoma in the first stage, and a comparison of the co-primary endpoints in the second randomized stage of the trial. Treatment will be divided into an 8-week induction and subsequent maintenance phases.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have signed and dated an Institutional Review Board/Independent Ethics Committee -approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal patient care
* Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study.
* All patients must be either Stage IIIb/c/d or Stage IV according to the American Joint Committee on Cancer (AJCC) (8th edition) and have histologically-confirmed melanoma that is felt to be surgically unresectable in order to be eligible. Please refer to the AJCC Cancer Staging Manual, 8th edition for a description of tumor, lymph node, metastasis and staging.

  * All melanomas, except ocular/uveal melanoma, regardless of primary site of disease will be allowed; mucosal melanomas are eligible.
  * Patients must not have received prior anticancer treatment for metastatic disease (for example, but not limited to, systemic, local, radiation, radiopharmaceutical).

oExceptions: Surgery for melanoma and/or post-resection brain radiotherapy (RT) if central nervous system (CNS) metastases and local radiation for locoregional disease and/or prior treatment with adjuvant nivolumab, dabrafenib and trametinib, pembrolizumab, interferon (IFN) or ipilimumab (IPI) (as described in Exclusion Criterion 8,4 full protocol below).

* All patients must have their disease status documented by a complete physical examination and imaging studies within 4 weeks prior to the first dose of study drug. Imaging studies must include computerized tomography (CT) scan of chest, abdomen, pelvis, and all known sites of resected disease in the setting of Stage IIIb/c/d or Stage IV disease, and brain magnetic resonance imaging ([MRI]; brain CT is allowable if MRI is contraindicated).
* Disease must be measurable by RECIST 1.1
* The complete set of baseline radiographic images must be available before treatment initiation.

Exclusion Criteria:

* Patients with untreated brain metastases, carcinomatosis meningitis or current ocular/uveal melanoma are excluded.
* Patients with previous non-melanoma malignancies are excluded unless a complete resection or remission was achieved at least 2 years prior to study entry and no additional therapy is required or anticipated to be required during the study period (exceptions include, but are not limited to, non-melanoma skin cancers, in situ bladder cancer, in situ gastric cancer or gastrointestinal stromal tumor, in situ colon cancers, in situ cervical cancers/dysplasia, or breast carcinoma in situ).
* Patients with active, known, or suspected autoimmune disease. Patients with type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll. For any cases of uncertainty, it is recommended that the Principal Investigator be consulted prior to signing informed consent.
* Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids are permitted in the absence of active autoimmune disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Number of Grades 3-5 Treatment-Related Immune-Related Adverse Events (irAE) per NCI CTCAE v 5.0 Criteria | week 24 (+/- 7 days)
  The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v 5.0) grades adverse events by the following scale:
  Grade 1 - Mild, Grade 2 - Moderate, Grade 3 - Severe, Grade 4 - Life-threatening, Grade 5 - Death
  Safety will be measured by physical examinations, vital sign measurements, Eastern Cooperative Oncology Group (ECOG) performance status evaluations, AE assessments, laboratory testing, electrocardiograms (ECGs), oxygen saturation, and concomitant medications.
Response Evaluation Criteria in Solid Tumors (RECIST 1.1) Category | week 24 (+/- 7 days)
  Each patient will be assigned one of the following categories:
  1. = Complete Response (CR) = Disappearance of all target lesions;
  2. = Partial Response (PR) = At least a 30% decrease in the sum of the longest diameter (LD) of target lesions.
  3. = Stable Disease (SD) = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD since treatment started.
  4. = Progressive Disease (PD) = At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
  5. = Early death from malignant disease
  6. = Early death from toxicity
  7. = early death because of other cause
  9 = Unknown (not assessable, insufficient data)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to Month 31
  Progression-Free Survival (PFS) will be reported as the time from first dosing to the first observation of disease progression or death due to any cause. If a patient has not progressed or died at the time of analysis, PFS will be censored on the date of the last disease assessment. Patients who do not have any tumor assessment on treatment will be censored on the day of the first dose.
Overall survival (OS) | Up to Month 31
  Overall Survival will be reported as the time from first dosing to death due to any cause. If a patient has not died at the time of analysis, OS will be censored as of their last known date alive (i.e., last time patient was contacted for any reason in the study). Patients who do not have any tumor assessment on treatment will be followed up for OS, and their date of death will be incorporated into the OS analysis.
Best overall response (iBOR) | week 24 (+/- 7 days)
  iBOR will be reported as the best timepoint response recorded from the time the measurement criteria are met for partial response (PR) or complete (CR), whichever is recorded first, until the date of documented PD or death.
Disease Control Rate (DCR) | Month 31
  Total number of patients whose best response outcome is a Complete Response (CR), Partial Response (PR) or Stable Disease (SD), divided by the total number of evaluable patients.
  Per Response Evaluation Criteria in Solid Tumors (RECIST v 1.1):
  CR = Disappearance of all target lesions; PR = At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; SD = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD since treatment started.
Duration of Overall Response | Month 31
  Among patients whose best response to treatment is a Complete Response (CR) or Partial Response (PR): The time between the date measurement criteria are met for PR or CR, whichever is recorded first, and the date of documented Progressive Disease (PD) or death.
  Per Response Evaluation Criteria in Solid Tumors (RECIST v 1.1):
  CR = Disappearance of all target lesions; PR = At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD PD = At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Duration of disease control | Up to Month 31
  Among patients who had an Overall Response Rate (ORR) outcome of Complete Response (CR), Partial Response (PR), or Stable Disease (SD): The time from first dosing to documented disease progression.
  Per Response Evaluation Criteria in Solid Tumors (RECIST v 1.1):
  CR = Disappearance of all target lesions; PR = At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; SD = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD since treatment started.
Immune-related Response Rate (irRR) per irRC criteria | Week 24
  The highest Immune-Related Response Criteria (irRC) designation given over 24 weeks, where:
  1. = Immune related complete response (irCR) = Complete disappearance of all tumor lesions
  2. = Immune related partial response (irPR) = A decrease relative to baseline of the immune related sum of products of diameters (irSPD) of 50% or greater
  3. = Immune related stable disease (irSD) = An evaluable response that fails to meet criteria for irCR or irPR, in the absence of progressive disease
  4. = Immune related progressive disease (irPD) = At least a 25% increase in the irSPD over the lowest irSPD
  5. = Immune related unknown response (irUN) = Tumor assessments that cannot be evaluated
Immune-related Response Rate (irRR) per irRC criteria | Month 31
  The total number of response-evaluable patients whose Immune Related Best Overall Response (irBOR) outcome is immune related complete response (irCR) or immune related partial response (irPR), per Immune-Related Response Criteria (irRC):
  irCR = Complete disappearance of all tumor lesions irPR = A decrease relative to baseline of the immune related sum of products of diameters (irSPD) of 50% or greater
Immune-related Disease Control Rate per irRC criteria | Month 31
  The total number of the response-evaluable patients whose Immune Related Best Overall Response (irBOR) outcome is immune related complete response (irCR), immune related partial response (irPR) or immune-related stable disease (irSD), per Immune-Related Response Criteria (irRC):
  irCR = Complete disappearance of all tumor lesions irPR = A decrease relative to baseline of the immune related sum of products of diameters (irSPD) of 50% or greater irSD = An evaluable response that fails to meet criteria for irCR or irPR, in the absence of progressive disease
Immune-related Progression-Free Survival (irPFS) | Month 31
  The time between first dosing and the date of immune-related progressive disease (irPD) or death, whichever occurs first. For patients with no recorded post-baseline tumor assessment, irPFS will be censored at the day of first dose. A patient who dies without reported irPD will be considered to have progressed on the date of death. For those who remain alive and have no irPD, irPFS will be censored on the date of last evaluable tumor assessment. Patients who do not have any tumor assessment on treatment will be censored on the day of the first dose.
  Per Immune-Related Response Criteria (irRC):
  irPD = At least a 25% increase in the irSPD over the lowest immune related sum of products of diameters
Duration of Immune-related Overall Response | Month 31
  Duration of Immune-related Overall Response will be computed for all patients whose irBOR outcome is either an irPR or irCR and is calculated from the time the measurement criteria are met for irPR or irCR, whichever is recorded first, until the date of documented PD or death by irRC
Duration of Immune-related Disease Control | Month 31
  Among patients with Immune-related Overall Response outcome of immune related complete response (irCR), immune related partial response (irPR), or immune-related stable disease (irSD): The time between the date treatment began and the date of documented disease progression.
  Per Immune-Related Response Criteria (irRC):
  irCR = Complete disappearance of all tumor lesions irPR = A decrease relative to baseline of the immune related sum of products of diameters (irSPD) of 50% or greater irSD = An evaluable response that fails to meet criteria for irCR or irPR, in the absence of progressive disease

CONTACTS AND LOCATIONS:
Overall Officials: Janice Mehnert, MD, Principal Investigator — NYU Langone Health
Locations (4):
- United States (4):
  - The Angeles Clinic at Cedars Sinai, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: No
Extensive correlative analyses will be performed using those samples, to be supported by RO1 funding applied for